CLINICAL TRIAL: NCT07326020
Title: Comparison of the Immediate Effects of Different Manual Therapy Methods in Physically Active Individuals With Pes Planus
Brief Title: Effectiveness of Manuel Therapy Methods in Pes Planus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hande Guney Deniz (Other)
Responsible Party: Sponsor-Investigator, Hande Guney Deniz, Prof. Dr., Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pesplanus2025
Record Dates: First submitted 2025-11-29; First posted 2026-01-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Pes Planus
Keywords: pes planus; manuel therapy; balance; range of motion; stiffness
MeSH Terms: conditions — Flatfoot | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention): healthy control group without intervention
- joint mobilization group (Experimental): subtalar and midtarsal joint mobilization in patients with flexible pes planus
  Interventions: Other: joint mobilization
- myofascial release group (Experimental): calf and plantar fascia release in patients with flexible pes planus
  Interventions: Other: myofascial release

INTERVENTIONS:
Other: joint mobilization — subtalar and midtarsal joint mobilization
  Arms: joint mobilization group
Other: myofascial release — calf and plantar fascia release
  Arms: myofascial release group

SUMMARY:
The aim of this study is to compare the immediate effects of joint-oriented manual therapy and soft tissue-oriented manual therapy on dorsiflexion angle, static and dynamic balance, muscle-tendon mechanical properties, and thermal variables in physically active individuals with flexible pes planus. The research will be conducted between November 2025 and January 2026 at Hacettepe University, Faculty of Physical Therapy and Rehabilitation. Individuals aged 18-35 years with a Tegner Activity Score between 4 and 6 will be included. Participants will be allocated into three groups: soft tissue-oriented manual therapy group, joint-oriented manual therapy group, and healthy control group. Following randomization, the respective intervention will be applied to the intervention groups, while no intervention will be administered to the control group. Assessments will include the dorsiflexion range of motion (weight-bearing lunge test), myotonometric measurements (Myoton-Pro), static balance (Kinvent force platform), dynamic balance (Y-balance test), and thermographic imaging (FLIR E52). The outcomes of this study are expected to contribute to understanding the immediate effectiveness of manual therapy approaches applied in asymptomatic pes planus and to identify the method providing optimal benefit. Furthermore, the differences observed between individuals with pes planus and healthy controls will serve as a guide for clinical assessments of pes planus.

ELIGIBILITY:
Inclusion Criteria for the Intervention Group:

* Navicular Drop Test ≥ 10 mm
* Foot Posture Index (FPI) > 6
* Tegner Activity Scale score between 4 and 6 (inclusive)
* Age between 18 and 35 years

Inclusion Criteria for the Control Group:

* Age between 18 and 35 years
* Navicular Drop Test < 10 mm
* Foot Posture Index (FPI) between 0 and 6 (inclusive)
* Tegner Activity Scale score between 4 and 6 (inclusive)

Exclusion Criteria for the Intervention Group:

* Diagnosis of posterior tibial tendinopathy by an orthopedic surgeon
* Presence of plantar fasciitis or moderate/severe hallux valgus
* History of lower extremity surgery or trauma
* Presence of neurological, metabolic, or other musculoskeletal disorders that may affect gait or balance performance
* Receipt of any treatment for pes planus within the past year
* Body mass index (BMI) greater than 30 kg/m²
* Regular participation in sports activities

Exclusion Criteria for the Control Group:

* Presence of plantar fasciitis or moderate/severe hallux valgus
* Presence of pes cavus deformity
* History of lower extremity surgery or trauma
* Presence of neurological, metabolic, or other musculoskeletal disorders that may affect gait or balance performance
* Body mass index (BMI) greater than 30 kg/m²
* Participation in professional-level sports activities

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2026-02-08 (Actual); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
static balance | 2 months
  1 Static Balance Measurement Static balance will be assessed using the Kinvent K-Plates (Kinvent, Montpellier, France), a reliable portable force plate with a 1000 Hz sampling rate. Participants will stand on one leg with hands on hips and the other leg flexed, focusing on a point 5 m away for 10 s. The test will be repeated with eyes closed. Postural oscillations (mm) and center of pressure (COP) (mm) data will be reported instantly via the mobile app. Each condition will be measured three times.
dynamic balance | 2 months
  Dynamic Balance Measurement Dynamic balance will be assessed using the Y-Balance Test platform (Move2Perform, Evansville, USA). Participants will reach in anterior, posteromedial, and posterolateral directions while maintaining single-leg stance, hands on hips. The maximum reach distance(cm) in each direction will be recorded. After practice trials, three valid attempts per direction will be completed. Results will be expressed as normalized composite scores(%) relative to limb length.

SECONDARY OUTCOMES:
myotonometric muscle tone | 2 months
  Muscle tone (Hz), will be assessed using the Myoton-Pro myotonometer (Myoton SA, Tallinn, Estonia; ICC: 0.76-0.86). Measurements will be taken from the Tibialis Anterior, Medial and Lateral Gastrocnemius, Soleus, Achilles tendon, and Plantar Fascia. The 3 mm probe will be applied perpendicularly to the skin (<3% error). Each site will be tested in standardized positions (supine or prone) and measured three times to obtain mean values for each mechanical property.
myotonometric muscle stiffness | 2 months
  Muscle stiffness (N/m) will be assessed using the Myoton-Pro myotonometer (Myoton SA, Tallinn, Estonia; ICC: 0.76-0.86). Measurements will be taken from the Tibialis Anterior, Medial and Lateral Gastrocnemius, Soleus, Achilles tendon, and Plantar Fascia. The 3 mm probe will be applied perpendicularly to the skin (<3% error). Each site will be tested in standardized positions (supine or prone) and measured three times to obtain mean values for each mechanical property.
ankle dorsiflexion range of motion | 2 months
  Ankle dorsiflexion ROM will be assessed with the Weight-Bearing Lunge Test (WBLT), a reliable method (ICC > 0.90). Participants will lunge toward a wall, keeping the heel in contact with the floor. The maximum distance (cm) from the great toe to the wall at which the knee touches without heel lift will be recorded. At this final position, a digital inclinometer will be placed on the tibia's midline to determine the tibial inclination angle (°). Measurements will be taken on both limbs under identical conditions.
skin surface thermographic measurement | 2 months
  Skin surface temperature (°C) will be assessed using a FLIR E52 thermographic camera (240×180 px infrared resolution, 50 mK sensitivity). Images will be captured in a controlled environment (23 ± 1°C; 40-60% humidity) and analyzed offline with Flir ResearchIR Max 4. Participants will acclimate for 15 min before testing. The emissivity will be set at 0.98, rainbow palette (27-35°C scale) applied, and the camera placed 1 m away, perpendicular to the skin. In the prone position, plantar fascia and sole temperatures will be recorded; in standing, calf and Achilles tendon regions will be imaged, with the highest temperature (°C) documented for each area.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Guney-Deniz, Prof. Dr, Study Director — Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Departmen of Musculoskeletal Physiotherapy and Rehabilitation, Ankara, Türkiye
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Will be shared with a plausible reason.
Supporting Information: Study Protocol, ICF